CLINICAL TRIAL: NCT02930603
Title: A Longitudinal Study of Function and Participation in Life Activities of Patients With Developmental Disabilities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-5441B
Record Dates: First submitted 2016-10-03; First posted 2016-10-12 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-01

CONDITIONS: Child Development Disorders
Keywords: Developmental Disabilities; Body function and body structure; Participation; Life activities; Quality of Life
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Control: Healthy child
- Experimental: Patients with Developmental Disabilities

SUMMARY:
A Longitudinal Study of Function and Participation in Life Activities of Patients with Developmental Disabilities

DETAILED DESCRIPTION:
Developmental Disabilities (DD) is defined as a group of neurodevelopmental issues, leading to significant lag in one or more areas (e.g. cognition, speech, motor, self-care and psychosocial function) for various reasons. On the basis of International Classification of Functioning, Disability and Health -Children and Youth Version (ICF-CY) framework, problems related to Developmental Disabilities further limit activities of daily living (ADL) and participation of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Developmental Disabilities
2. Age 0-25 y/o
3. Agree to sign informed consent

Exclusion Criteria:

1. Active medical condition (e.g. infection)
2. Concurrent progressive or degenerative disease (e.g. neurogenerative disease)
3. Concurrent illness or disease not typically associated with DD (e.g. pneumonia)

Ages: 7 Days to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Control and experimental groups
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-04; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of general developmental for Healthy child and patients with Developmental Disabilities in 6 months and 12 months | baseline, 6 months, 12 months
  Comprehensive Developmental Inventory for Infants and Toddlers
Change from baseline of body function & structures in 6 months and 12 months | baseline, 6 months, 12 months
  Bruininks- Oseretsky Test of Motor Proficiency II
Change from baseline of upper extremity function & structures in 6 months and 12 months | baseline, 6 months, 12 months
  Quality of upper extremity skills test
Change from baseline of lower extremity function & structures in 6 months and 12 months | baseline, 6 months, 12 months
  Pediatric Balance Scale
Change from baseline of Sensory and Perceptual function in 6 months and 12 months | baseline, 6 months, 12 months
  Sensory Profile

SECONDARY OUTCOMES:
Change from baseline of activities in 6 months and 12 months | baseline, 6 months, 12 months
  Functional Independence Measure for Children
Change from baseline of Participation in 6 months and 12 months | baseline, 6 months, 12 months
  Children Assessment of Participation and Enjoyment, Preferences for Activity of Children
Change from baseline of Quality of Life in 6 months and 12 months | baseline, 6 months, 12 months
  TNO-AZL Child Quality of Life Questionnaire
Change from baseline of Personal & Environment factor in 6 months and 12 months | baseline, 6 months, 12 months
  Parenting Stress Index,
Change from baseline of Rehabilitation & community service factor in 6 months and 12 months | baseline, 6 months, 12 months
  Measure of Processes of Care

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No